CLINICAL TRIAL: NCT06759779
Title: Effects of Inspiratory and Expiratory Muscle Strength Training on Respiratory Functions and Performance in Adolescent Volleyball Players
Brief Title: Inspiratory and Expiratory Muscle Training in Adolescent Volleyball Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeliha ÇELİK, Asst.Prof, Amasya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 474032
Record Dates: First submitted 2024-12-13; First posted 2025-01-06 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Adolescent Development
Keywords: pulmonary functions; muscle training; adolescent health; volleyball players

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inspiratory muscle training group (Experimental)
  Interventions: Device: inspiratory muscle training
- expiratory muscle training group (Experimental)
  Interventions: Device: expiratory muscle training

INTERVENTIONS:
Device: inspiratory muscle training — Inspiratory muscle training will be performed
  Arms: inspiratory muscle training group
Device: expiratory muscle training — Expiratory muscle training will be performed
  Arms: expiratory muscle training group

SUMMARY:
This study will investigate the effects of inspiratory and expiratory muscle training on respiratory muscle strength, pulmonary function, and performance status in adolescent athletes

DETAILED DESCRIPTION:
In the literature, it has been shown in a limited number of studies that respiratory muscle training in sports such as football, cycling, swimming, and rugby reduces athletes' perceived exertion levels. However, the effects of inspiratory and expiratory muscle training on respiratory muscle strength, pulmonary function, and performance status in adolescent athletes are still unclear. Therefore, this study has been planned.

ELIGIBILITY:
Inclusion Criteria:

* Athletes aged 12-18 who train at a submaximal level at least 3 days a week

Exclusion Criteria:

* Adolescents with any history of chronic lung disease
* unable to comply with the test and training
* unwilling to participate in the study

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | First day
  Maximal inspiratory and expiratory muscle strength will be evaluated using mouth pressure device .

SECONDARY OUTCOMES:
Constant load-inspiratory muscle endurance test | First day
  It will be evaluated with inspiratory muscle trainer
FEV1 | First day
  ulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respratory Society criteria. FEV1 will be evaluated. The percentage of predicted value <70% will be expressed as abnormal
FVC | First day
  ulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respratory Society criteria. FEV1 will be evaluated. The percentage of predicted value <70% will be expressed as abnormal
FEV1/FVC | First day
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respratory Society criteria. FEV1/FVC will be evaluated.
PEF | First day
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respratory Society criteria. PEF will be evaluated. The percentage of predicted value <70% will be expressed as abnormal
FEF2575 | First day
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respratory Society criteria. FEF2575 will be evaluated. The percentage of predicted value <50% will be expressed as abnormal
Athletic performance | second day
  Performance will be evaluated with shuttle run test
Fat free mass Body compositions | second day
  Fat free mass (kg) will be evaluated with bioelectrical impedance analyzer
Fat mass Body compositions | second day
  Fat mass (kg) will be evaluated with bioelectrical impedance analyzer
Fat percentage Body compositions | second day
  Fat percentage (%) will be evaluated with bioelectrical impedance analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Emek, Turkey (Türkiye)